CLINICAL TRIAL: NCT03278158
Title: A Single-dose Dose Escalation Trial in a Randomised, Single-blind, Placebo-controlled Group-comparison Design to Investigate the Safety and Tolerability of XEN-D0501 in Patients With Diabetes Mellitus Type 2
Brief Title: A Single-dose Trial to Investigate the Safety and Tolerability of XEN-D0501 in Patients With Diabetes Mellitus Type 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pila Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PP-CT01
Record Dates: First submitted 2017-08-28; First posted 2017-09-11 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: safety; tolerability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Each subject will be randomised to one of four treatments, placebo and three different single oral doses of XEN-D0501. Cohorts of 8 patients are run subsequently where of 2 patients receive placebo and 6 patients receive XEN-D0501 beginning with the 1 mg dose followed by the 2, 4 and 8 mg dose groups. Each treatment step will be completed consecutively and progression to next dose level depend on good safety and tolerability on the previous dose level.
Who Masked: Participant
Masking Description: The type of treatment is blinded for the subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive a single oral tablet containing no active drug.
  Interventions: Drug: Placebo
- XEN-D0501, 1 mg/tablet (Experimental): Subjects in this arm will receive a single oral tablet of XEN-D0501, 1 mg/tablet
  Interventions: Drug: XEN-D0501, 1 mg/tablet
- XEN-D0501, 2 mg/tablet (Experimental): Subjects in this arm will receive a single oral tablet of XEN-D0501, 2 mg/tablet. Discontinued after 2 patients due to good safety. Escalation to higher dose levels in whole study (1, 2 and 4 mg changed to 1, 4 and 8 mg)
  Interventions: Drug: XEN-D0501, 2 mg/tablet
- XEN-D0501, 4 mg/tablet (Experimental): Subjects in this arm will receive a single oral tablet of XEN-D0501, 4 mg/tablet
  Interventions: Drug: XEN-D0501, 4 mg/tablet
- XEN-D0501, 8 mg/tablet (Experimental): Subjects in this arm will receive a single oral tablet of XEN-D0501, 8 mg/tablet
  Interventions: Drug: XEN-D0501, 8 mg/tablet

INTERVENTIONS:
Drug: Placebo — Subjects in the placebo arm will receive a single oral tablet containing no active drug.
  Arms: Placebo
Drug: XEN-D0501, 1 mg/tablet — Subjects in this arm will receive a single oral tablet of XEN-D0501, 1 mg/tablet
  Arms: XEN-D0501, 1 mg/tablet
Drug: XEN-D0501, 2 mg/tablet — Subjects in this arm will receive a single oral tablet of XEN-D0501, 2 mg/tablet
  Arms: XEN-D0501, 2 mg/tablet
Drug: XEN-D0501, 4 mg/tablet — Subjects in this arm will receive a single oral tablet of XEN-D0501, 4 mg/tablet
  Arms: XEN-D0501, 4 mg/tablet
Drug: XEN-D0501, 8 mg/tablet — Subjects in this arm will receive a single oral tablet of XEN-D0501, 8 mg/tablet
  Arms: XEN-D0501, 8 mg/tablet

SUMMARY:
This is a single-dose dose escalation trial in a randomised, single-blind, placebo-controlled group-comparison design to investigate the safety and tolerability of XEN-D0501 in subjects with diabetes mellitus type 2 where life style changes and treatment with metformin has failed to effectively reduce blood glucose concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must give his/her signed and dated informed consent before any trial-related activities. Trial-related activities are any procedures that would not have been performed during the normal management of the subject.
2. Diagnosis of type 2 diabetes mellitus
3. In treatment with metformin, but no other anti-diabetic drugs
4. In treatment with an ACE-inhibitor but no other anti-hypertensive drugs
5. HbA1C (glycosylated haemoglobin A1C) 6.5-10 %
6. Age between 30 and 70 years (both inclusive).

Exclusion Criteria:

1. A subject with a history of significant multiple drug allergies or with a known or suspected allergy to the trial product or any medicine chemically related to the trial product, as judged by the Investigator.
2. A subject who has a supine blood pressure at screening (including those on anti-hypertensives), after resting for 5 min, outside the range of 90-140 mmHg systolic or 50-90 mmHg diastolic (excluding white-coat hypertension; therefore, if a repeated measurement on a second screening visit shows values within the range, the subject can be included in the trial).
3. A subject who is in pharmacological treatment of hypertension if the current treatment includes other than an ACE-inhibitor
4. A subject who has a clinically significant abnormal ECG at screening, as judged by the investigator.
5. A subject who has participated in any other trials involving investigational products within the 3 months preceding the start of dosing.
6. A subject who has donated any blood or plasma in the past month or in excess of 500 mL within the 3 months preceding screening.
7. A subject who has a significant history of alcoholism or drug/chemical abuse as per investigator's judgement, or who has a positive result in the urine drug/alcohol screen at screening visit.
8. A subject who smokes more than 5 cigarettes, or the equivalent, per day and is unable to refrain from smoking during the in-house periods as determined by the Investigator.
9. A subject with mental incapacity or language barriers which preclude adequate understanding or cooperation, who is unwilling to participate in the trial, or who in the opinion of their general practitioner or the Investigator should not participate in the trial.
10. Surgery or trauma with significant blood loss within the last 2 months prior to dosing.
11. A subject with a history of or presence of cancer, or any clinically significant, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (with the exception of diabetes mellitus type 2 and euthyroid struma), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders.
12. Cardiac problems defined as: decompensated heart failure (New York Heart Association (NYHA) class III and IV) at any time and/or angina pectoris and/or acute myocardial infarction within the last 12 months.
13. A subject with a clinically significant abnormal haematology or biochemistry tests at screening visit, as judged by the Investigator considering the underlying disease.
14. Current treatment with drugs known to interfere with glucose metabolism such as systemic corticoids and monoamine oxidase inhibitors (MAO) inhibitors.
15. A subject who has proliferative retinopathy or maculopathy, and/or severe neuropathy, in particular autonomic neuropathy, as judged by the Investigator.
16. Haemoglobin < 6.2 mmol/l, total leukocyte count < 3.0 x 109/l, thrombocytes <100 x 109/l, serum creatinine levels ≥ 126 µmol/l (male) or ≥ 111 µmol/l (female), bilirubin > 3 x ULN, alanine aminotransferase > 2 x the upper limit of normal (ULN), alkaline phosphatase > 2 x ULN, one re-test within a week is permitted.
17. Previous participation (randomisation) in this trial.
18. Any condition that would interfere with trial participation or evaluation of results, as judged by the investigator and/or sponsor
19. Recurrent major hypoglycaemia or hypoglycaemic unawareness, as judged by the Investigator.
20. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (Adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral hormonal contraceptives (p-pills), implantants, transdermal patches, p-ring or depot injection, sexual abstinence or vasectomised partner). A male subject who is sexually active and has not been surgically sterilised must be informed that he must ensure that his partner practices effective contraception, as stated above, or he must refrain from sexual intercourse during the trial and until 90 days after completion of the trial. This is to prevent the possibility of a pregnancy from spermatocytes that can potentially be damaged by trial medication.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single ascending oral doses of XEN-D0501, (1, 2, 4 and 8 mg) versus placebo in type 2 diabetic patients in treatment with metformin (Incidence of adverse events in type 2 diabetic patients) | 1-3 weeks
  Incidence of adverse events in type 2 diabetic patients

CONTACTS AND LOCATIONS:
Overall Officials: Henning Beck-Nielsen, Dr., Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No